CLINICAL TRIAL: NCT02763488
Title: Blood Flow Restriction Training Following Primary Total Knee Arthroplasty
Brief Title: Blood Flow Restriction Training Following Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Tennent, Orthopaedic Surgery Resident, San Antonio Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2016.109
Record Dates: First submitted 2016-05-02; First posted 2016-05-05 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis
Keywords: blood flow restriction training; occlusion training; total knee arthroplasty; post-operative rehabilitation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard physical therapy (Active Comparator): These individuals will conduct physical therapy for 12 sessions as per the institutional standard physical therapy protocol
  Interventions: Other: Standard physical therapy
- Blood flow restriction (Experimental): These individuals will conduct physical therapy for 12 sessions with the addition of blood flow restriction interventions to their standard physical therapy
  Interventions: Device: DelfiPTS tourniquet system

INTERVENTIONS:
Device: DelfiPTS tourniquet system
  Arms: Blood flow restriction
Other: Standard physical therapy
  Arms: Standard physical therapy

SUMMARY:
This study will evaluate blood flow restriction training as a rehabilitation modalities following total knee arthroplasty in order to determine if patient reported outcomes and objective functional outcomes can be improved through post-operative rehabilitation compared to standard physical therapy modalities currently in use.

DETAILED DESCRIPTION:
Patients will be enrolled preoperatively in order to measure preoperative functional measures. They will then be followed at predetermined intervals post-operatively. All subjects will begin the study related physical therapy 6 weeks post-operatively and continue for 12 sessions. At the conclusion of 12 sessions, subjects will be retested to determine improvement. Subjects will then be followed for two years post-operative.

ELIGIBILITY:
Inclusion Criteria:

* S/p primary Total Knee Arthroplasty and cleared by surgeon for continued physical therapy
* Males and females 50-79 years of age
* Ability to consent to study enrollment
* Able to participate fully in physical therapy
* Tricare Beneficiary
* Implant restricted: primary cruciate retaining or posterior stabilized total knee arthroplasty
* Knee range of motion of surgical extremity from a minimum of 5 degrees from full extension to 90 degrees of flexion**

  * only screened at secondary screening

Exclusion Criteria:

* Unable to consent for study participation
* Unable to participate in preoperative testing
* Any ligamentous or bony reconstruction performed at time of surgery that limits weight bearing or rehabilitation protocol
* History of deep venous thrombosis
* Injury or recent procedure to contralateral extremity within past 6 months
* History of endothelial dysfunction
* History of Peripheral Vascular Disease
* Patient endorsement of easy bruising
* Revision Total Knee Arthroplasty
* History of Surgical wound complication on involved extremity
* History of Cerebral Vascular Event
* History of Dementia
* History of Neuromuscular disorder
* History of Chronic Obstructive Pulmonary Disease requiring oxygen supplementation or limiting participants ability to perform therapy and/or testing
* History of previous intra-articular fracture of surgical extremity requiring open reduction and internal fixation or external fixation
* History of Sickle cell trait and/or disease
* Previously participated in blood flow restriction training interventions
* Planned or unplanned additional surgical procedures affecting their ability to complete all session of physical therapy or testing during the following 6 months from their primary intervention
* Patient reported history of functionally limiting arthritis in non-surgical lower extremity or ipsilateral hip or ankle
* History or previous contralateral total knee arthroplasty
* Any history of previous total hip arthroplasty

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
quadriceps strength | baseline up to 2 years post operative
  quadriceps strength via dynamometer

SECONDARY OUTCOMES:
Patient reported outcome 1: KOOS | baseline up to 2 years post operative
  Patient reported measure of subject pain and function
Patient reported outcome 2: PROMIS Global Health | baseline up to 2 years post operative
  PROMIS Global Health is a global measure of mental and physical health
Patient reported outcome 3: Promis-29 | baseline up to 2 years post operative
  NIH validated patient reported outcome measure evaluating multiple mental and physical domains
Patient reported outcome 4: Pain Visual analog score | baseline up to 2 years post operative
  Patient pain rating
Physical Outcome measure 1: Four square step test | baseline up to 2 years post operative
  Validated functional outcome evaluating lower extremity function
Physical Outcome measure 2: Sit to stand test | baseline up to 2 years post operative
  Validated functional outcome evaluating lower extremity function
Physical Outcome measure 3: 6 minute walk test | baseline up to 2 years post operative
  Validated functional outcome evaluating lower extremity function
Physical Outcome measure 4: Timed up and go test | baseline up to 2 years post operative
  Validated functional outcome evaluating lower extremity function
Physical Outcome measure 5: Timed stair ascent | baseline up to 2 years post operative
  Validated functional outcome evaluating lower extremity function

CONTACTS AND LOCATIONS:
Overall Officials: David J Tennent, MD, Principal Investigator — San Antonio Military Medical Center
Locations (1):
- San Antonio Military Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No